## [LOCAL LOGO]



| CONSENT FORM | | | |
|---|---|---|---|
| Full Trial Title | Longitudinal Asse | essment of Multip | ole Organs in Patients with Type 2 Diabetes (MODIFY) |
| Site ID Code | MOD-XXX | Participant ID | |
| Principal<br>Investigator | Principal Investigator | | |

This form outlines what you agree to when you decide to participate in the above research study. All study information is provided in the patient information sheet and will have been shared and discussed with you in advance of completion of this form.

| | | Please initial relevant box |
|---|---|---|
| 1. | I confirm that I have read and understood the information sheet dated 03 February 2022, version 6.0 for the above research study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw from the study at any time without any given reason and without my medical or legal rights being affected. | |
| 3. | I understand that collected images, samples and associated data will be used by the Study Investigators for the purposes of this study. | |
| 4. | I understand that my medical notes will be consulted during my active participation in the study and afterwards at 1, 3 and 5 years from my first visit. I give permission for the study team to access my medical records in order to obtain health outcome data related to diabetes and associated complications for the full duration of the study. | |
| 5. | I understand that relevant sections of medical notes and data collected during the study may be looked at by individuals from Perspectum, and from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my data. | |
| 6. | I understand that the information and data collected about me may be used in an anonymous format to support other research by the study team in the future, including for research and development of MRI technology by Perspectum. It will not be possible for me to be identified from this information. | |
| 7. | I understand that the MRI scans performed in this study are exclusively for research purposes and are not used for medical diagnosis. If a concern is raised about a possible finding on my scan, it will be discussed with a relevant specialist and I will be contacted directly. | |
| 8. | In the case that an incidental finding is discovered on my research MRI, I give permission for the team to contact and inform my GP. | |
| 9. | I agree for my GP to be informed about my participation in this study. | |
| 10. | I agree to take part in this research study. | |

Subject:
Principal Investigator:
Short Title:

| Informed Consent Form |
|-------------------------|
| Princiipal Investigator |
| MODIFY |

264182 03Feb2022, v4.0 1 of 2

Version/Date: Page:

IRAS ID:

## [LOCAL LOGO]



| 11. | [OPTIONAL] I give permission for the storage of small amounts of blood or parts of cells, including genetic material, for analysis at a later date by the study team. I understand that the samples will be stored with a unique study code that will not provide any identifying information about me. | Yes | No |
|---|---|---|---|
| 12. | [OPTIONAL] I give permission for the study team to provide tissue samples to the NIHR National Biosample Centre ahead of future testing by the study team. I understand that this information will be stored in a database with a unique study code that will not provide any identifying information about me. | Yes | No |
| 13. | [OPTIONAL] I agree to have an echocardiogram during this study. | Yes | No |
| 14. | [OPTIONAL] I understand that the echocardiogram scans performed in this study are exclusively for research purposes and are not used for medical diagnosis. If a concern is raised about a possible finding on my scan, it will be discussed with a relevant specialist and you will be contacted directly. In the case that an incidental finding is discovered on my research echocardiogram, I give permission for the team to contact and inform my GP. | Yes | No |
| 15. | [OPTIONAL] I agree for my samples to be used in future ethically approved research, here or abroad. | Yes | No |
| 16. | [OPTIONAL] I agree to be contacted by Perspectum about future research activities in which I may be interested. I understand that agreeing to be contacted does not oblige me to participate in any further investigations. I agree for Perspectum to retain my study data, which can be linked to my contact details to identify studies specifically suited to my health status. I understand that my contact details will be stored in a dedicated, secure database with restricted access. | Yes | No |
| 17. | If YES to [16] please provide a contact telephone number and/or email address: | | |
| | Name ( <i>Please Print</i> ): | | |
| | Telephone: | | |
| | Email: | | |
| Name | e of Participant Date Signature | | |
| Name | e of Person Taking Consent Date Signature | | |
| | Subject: Informed Consent Form IRAS ID: 264182 | | |

Subject:
Principal Investigator:
Short Title:

| Informed Consent Form | IRAS ID: |
|-------------------------|---------------|
| Princiipal Investigator | Version/Date: |
| MODIFY | Page: |

| 264182 |
|-----------------|
| 03Feb2022, v4.0 |
| 2 of 2 |